CLINICAL TRIAL: NCT01187082
Title: A Clinical, Randomized, Comparative, Non-blinded Study on the Effect of Bladdertraining in Groups Compared to Individual Bladdertraining for Female Patients With Overactive Bladder.
Brief Title: Grouptraining for Overactive Bladder in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BLATRA 01
Record Dates: First submitted 2010-08-10; First posted 2010-08-23 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2011-02

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; women; bladder training; groups
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bladdertraining group (Experimental): Cognitive training in groups at hospital by a continence nurse in 3 sessions (1 hour)over a period of 1 month. Follow up after 1 month. During all 2 month the patient has selfinitiatied daily training with a pocket bladder schedule.
  Interventions: Behavioral: bladdertraining in groups
- bladdertraining individually (Active Comparator): Cognitive training individually at hospital by a continence nurse in 3 sessions (1 hour)over a period of 1 month. Follow up after 1 month. During all 2 month the patient has selfinitiatied daily training with a pocket bladder schedule.
  Interventions: Behavioral: bladdertraining individually

INTERVENTIONS:
Behavioral: bladdertraining in groups — Cognitive training in groups of 4 patients at hospital by a continence nurse in 3 sessions (1 hour)over a period of 1 month. Follow up after 1 month. During all 2 month the patient has selfinitiatied daily training with a pocket bladder schedule.
  Arms: bladdertraining group
Behavioral: bladdertraining individually — Cognitive training individually at hospital by a continence nurse in 3 sessions (1 hour)over a period of 1 month. Follow up after 1 month. During all 2 month the patient has selfinitiatied daily training with a pocket bladder schedule.
  Arms: bladdertraining individually

SUMMARY:
Hypothesis:the effect of bladdertraining in groups for patients with OAB (overactive bladder syndrome) equals the effect of bladdertraining individually for patients with overactive bladder.

The effect of the training is measured in a 3 dimensional scope by the means of 3 primary outcome measures used in the statistical evaluation. Symptoms of OAB (either (1)urgencyepisodes or (2)urgencyincontinence) and (3)quality of life (VAS score).

DETAILED DESCRIPTION:
Program consisting of 3 hourly sessions with bladdertraining and daily training with a pocket bladder schedule. patients are randomised either for groups or individual training with a continence nurse over a period of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* women at the age of 18 and more
* patients with overactive bladder

Exclusion Criteria:

* dominance of stress incontinence
* not able to attend sessions
* do not to understand danish
* do not want training in groups or individual
* hormonebalanced (if postmenopausal with added hormonetreatment for at least 2 months)
* no treatment for OAB up till 1 month before study and during study
* no renal or neurological diseases, symptomatic cystitis or non regulated diabetes
* no pregnancy during study
* no normal gynecological examination
* no operation in pelvis up till 3 month before studystart
* no polyuria measured 2 times before studystart (> 40 ml/ kg/ day)
* no upstart of treatment with medication during studystart which according to the investigator can create symptoms of OAB
* no participation in other CT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
urgencyepisodes | after 2 month (end of study)
  with a bladderdiary episodes are counted at studystart / after 3 sessions of training and after 2 month (studyend)
urgeincontinence | after 2 month (studyend)
  with a bladderdiary episodes are counted at studystart / after 3 sessions of training and after 2 month (studyend)
VAS score from ICI_OAB_Q | after 2 month (studyend)
  with the ICI_OAB_Q counted before studystart / after 3 sessions/ after 2 month (studyend)

SECONDARY OUTCOMES:
voiding frequency | after 2 month (studyend)
  counted from a bladder diary before studystart/ after 3 sessions of training/ after 2 month (studyend)
Compliance in training | after 2 month (studyend)
  counted from a pocket bladder schedule at every training session (3 times)and after 2 month (studyend)
Adverse events | after 2 month (studyend)
  asked at every training session (3 times)and after 2 month (studyend). Patients are supposed to report in if any AEs during study

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Kaysen, nurse, Principal Investigator — Århus Universitetshospital, Skejby
Locations (5):
- Denmark (5):
  - Århus Universitetshospital, Skejby, urogynaekology dep., Aarhus
  - Glostrup Hospital, Glostrup Municipality
  - Kolding Sygehus, urogynecology department, Kolding
  - Sønderborg Sygehus, Gynækologiske Ambulatorium, Sønderborg
  - Regionshospitalet Viborg, Kontinensklinikken, Viborg

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598